CLINICAL TRIAL: NCT01458509
Title: A Comparison of the Feasibility and Psychometric Properties of Paper vs. Web vs. Automated Telephone Administration of Patient Reported Outcome Surveys
Brief Title: Feasibility and Psychometric Properties of Paper vs. Web vs. Automated Telephone Administration of Patient Reported Outcome Surveys
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-101
Record Dates: First submitted 2011-10-18; First posted 2011-10-25 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Quality of Life; patient outcomes; questionaires; 11-101
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- IVRS ( interactive voice response system) EASP: Telephone Group with Nurse Intervention
  Interventions: Behavioral: surveys
- Web EASP: Web Group with Nurse Intervention
  Interventions: Behavioral: surveys
- IVRS ( interactive voice response system) No EASP: Telephone Group without nurse intervention
  Interventions: Behavioral: surveys
- Web No EASP: Web Group without nurse intervention
  Interventions: Behavioral: Surveys

INTERVENTIONS:
Behavioral: surveys — IVRS: An interactive voice response system (IVRS) is an automated telephone platform. The IVRS system will allow the participant to complete the survey when they receive the call and/or to call the system within the survey window to complete the survey. In each group, administration of a survey including the BFI, PRO-CTCAE sexual function items, and QOL LASA and in each group, the survey will be conducted once a month over a six-month period. The intervention will be an email alert to study personnel (EASP). Patients randomized to EASP will receive a phone call if their bowel function by the clinical office nurse if the study personnel determine that the patient's BFI, as reported on the monthly survey, is less than 53 (lowest quartile scores). Interventions that may occur include dietary and/or medication advice at the discretion of the office staff.
  Groups: IVRS ( interactive voice response system) EASP
Behavioral: surveys — Web: Study participants will be sent an email containing a link to the web survey. The participants will click on the link and complete the survey. Study participants may also login to the web survey independent of the link received via email. In each group, administration of a survey including the BFI, PRO-CTCAE sexual function items, and QOL LASA and in each group, the survey will be conducted once a month over a six-month period. Patients randomized to EASP will receive a phone call if their bowel function by the clinical office nurse if the study personnel determine that the patient's BFI, as reported on the monthly survey, is less than 53 (lowest quartile scores). Interventions that may occur include dietary and/or medication advice at the discretion of the office staff.
  Groups: Web EASP
Behavioral: surveys — IVRS: An interactive voice response system (IVRS) is an automated telephone platform. The IVRS system will allow the participant to complete the survey when they receive the call and/or to call the system within the survey window to complete the survey. In each group, administration of a survey including the BFI, PRO-CTCAE sexual function items, and QOL LASA and in each group, the survey will be conducted once a month over a six-month period. This group will not get a phone call.
  Groups: IVRS ( interactive voice response system) No EASP
Behavioral: Surveys — Web: Study participants will be sent an email containing a link to the web survey. The participants will click on the link and complete the survey. Study participants may also login to the web survey independent of the link received via email. In each group, administration of a survey including the BFI, PRO-CTCAE sexual function items, and QOL LASA and in each group, the survey will be conducted once a month over a six-month period. This group will not receive a phone call.
  Groups: Web No EASP

SUMMARY:
It can be difficult to obtain the perspective of patients who have had bowel surgery. This study is being done because the investigators are trying to find out whether patient-reported outcomes, (results reported to investigators by the patient), on a regular basis, will help the investigators provide better patient care and symptom management.

Therefore, the purpose of this study is to determine if it is possible and if it is useful to their medical care for patients who have had bowel surgery to complete surveys about their symptoms on a regular basis. In this study the surveys are completed from home, by web or by telephone, every month for 6 months. The results of this study will guide the design of large research studies on cancer-related bowel function.

The purpose of this study is to develop a bowel function questionnaire for patients with colorectal cancer. The questionnaire will be used in future clinical trials to assess bowel function.

ELIGIBILITY:
Inclusion Criteria:

Aim 1:

* Stage I-III rectal cancer
* Post sphincter preserving surgery with restoration of bowel continuity within last 4-6 weeks at MSKCC.
* Access to web and email from home
* Web avidity (≥2 uses of email/week)
* Able to read and write in English
* Age ≥ 18

Aim 2:

* Stage I-III colon and rectal cancer
* Post surgical resection of primary tumor at MSKCC
* Access to web and email from home
* Web avidity (≥2 uses of email/week)
* Able to read and write in English
* Age ≥ 18

Exclusion Criteria:

Aim 1:

* Metastatic disease - Auditory, visual or motor impairment that would preclude ability to use telephone and/or computer.
* Stoma
* Participated in Aim 2
* Definitive SPS = Transanal Excision (TAE) or Transanal Endoscopic Microsurgery (TEM)

Aim 2:

* Metastatic disease - Auditory, visual or motor impairment that would preclude ability to use telephone and/or computer.
* Stoma
* Participated in Aim 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be screened in colorectal surgery clinics on the 3rd floor of the MSKCC 53rd Street outpatient clinic buildings or at the Main Hospital at 1275 York Avenue or while they are an inpatients. Patients will be approached within 1-5 weeks post operatively to ensure that they can complete the first survey within the 4-6 week window.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2011-10-11 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
clinically useful to collect patient-reported data | 6 months
  using electronic methods (interactive voice response system (IVRS) or web interface)
feasibility of electronic PRO assessment | 2 years
  we define feasibility as being the completion of 4/6 surveys. A complete survey is defined as having responses to 17/24 items (70%) on the survey. The administration mode will be deemed feasible if >=70% of patients complete 4/6 surveys.

SECONDARY OUTCOMES:
psychometric equivalence | 2 years
  Relevant in colorectal cancer trials via three different modes of administration: Web, IVRS, paper. The primary interest is the psychometric properties of the total score and subscale scores of the BFI, however individual items scores will be examined as well.
problems people experience | 2 years
  With bowel function, bladder function, and sexual function over the course of treatment for rectal cancer and to identify the types of information that would be helpful to future patients. Patients who were enrolled in Aim 1 will be asked to participate in a 30-45 minute telephone interview. A total of 20 interviews will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Garcia-Aguilar, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm